CLINICAL TRIAL: NCT04287920
Title: A Phase II Study Evaluating the Safety of Acamprosate for Alcohol Use Disorder in Alcohol-related Liver Disease
Brief Title: Acamprosate Safe to Use in Individuals With Liver Disease.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Douglas (Doug) A. Simonetto, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 18-010902
Record Dates: First submitted 2020-01-31; First posted 2020-02-27 (Actual); Results first posted 2022-12-20 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-11

CONDITIONS: Alcohol-related Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alcohol-related liver disease and AUD, MELD-NA less than 20 (Experimental): The first 5 patients enrolled = AUD (alcohol use disorder) w/MELD-Na (model for end stage liver disease sodium) score less than 20.
  Interventions: Drug: Acomprosate
- Alcohol-related liver disease and AUD, MELD-NA more than 20 (Experimental): The second 5 patients enrolled = AUD (alcohol use disorder) w/MELD-Na (model for end stage liver disease sodium) score more than 20.
  Interventions: Drug: Acomprosate

INTERVENTIONS:
Drug: Acomprosate — Acamprosate will be administered orally and will be dosed at 333 mg three times a day, if tolerated it will be increased to 666 mg three times a day. Acamprosate will be administered for a total of 3 months

SUMMARY:
Is acamprosate safe to use in individuals with liver disease.

DETAILED DESCRIPTION:
Adult patients aged 21 or over with a diagnosis of alcohol-related liver disease and alcohol use disorder (AUD) and abstinent from alcohol for at least 2 weeks (but not more than 6 months) prior to initiating acamprosate treatment.

ELIGIBILITY:
Inclusion criteria:

* Aged 21 or over
* Diagnosis of alcohol-related liver disease and AUD.

  * The diagnosis of alcohol-related liver disease will be determined by a hepatologist based on history of regular and excessive alcohol consumption in the absence of other causes of liver cirrhosis or acute hepatitis, compatible clinical, imaging and laboratory findings and typical histology on liver biopsy, if performed. Underlying liver disease may include alcoholic hepatitis, advanced (F3-F4) fibrosis, and/or portal hypertension.
  * The diagnosis of AUD will be determined by a hepatologist and/or addiction psychiatrist based on history obtained that is consistent with DSM-5 diagnostic criteria for AUD (all categories of mild, moderate and severe considered eligible) (American Psychiatric Association, 2013; questions from NIH, 2016).
* Abstinent from alcohol for at least 2 weeks (but not more than 6 months) prior to initiating acamprosate treatment.
* At study enrollment, initial MELD-Na score must be less than 20 for the five individuals enrolling in the first phase of the pilot safety assessment. The second phase of the pilot safety assessment will include individuals with a MELD-Na of 20 or more at enrollment.
* Have capacity to provide consent themselves

Exclusion criteria:

* Individuals with a glomerular filtration rate (GFR) of less than 30 ml/min
* Congestive heart failure (NYHA class II or higher)
* Hypotension, requiring the use of vasoconstrictors (i.e. midodrine)
* Pregnancy, lactation or refusal to use a reliable method of birth control if a sexually active female of childbearing potential. Although no human trial data is available, animal studies suggest possible teratogenic effects of acamprosate (Merck, 2005).

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2022-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas A Simonetto, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu T, Mousa OY, Kulai T, Larson C, Olofson A, Kamath PS, Shah VH, Taner T, Sanchez W, Simonetto DA. Safety of Acamprosate in Patients With Alcohol-Associated Liver Disease: A Single-Arm Phase 2 Trial. Mayo Clin Proc. 2025 Jun;100(6):954-961. doi: 10.1016/j.mayocp.2024.12.013. Epub 2025 Mar 26. PMID 40136257
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Alcohol-related Liver Disease and AUD, MELD-NA Less Than 20: The first 5 patients enrolled = AUD (alcohol use disorder) w/MELD-Na (model for end stage liver disease sodium) score less than 20.
  Acamprosate: Acamprosate was administered orally and was dosed at 333 mg three times a day, if tolerated it was increased to 666 mg three times a day. Acamprosate was administered for a total of 3 months
- Alcohol-related Liver Disease and AUD, MELD-NA More Than 20: The second 5 patients enrolled = AUD (alcohol use disorder) w/MELD-Na (model for end stage liver disease sodium) score more than 20.
  Acamprosate: Acamprosate was administered orally and was dosed at 333 mg three times a day, if tolerated it was increased to 666 mg three times a day. Acamprosate was administered for a total of 3 months
Period: Overall Study
Arm/Group | Alcohol-related Liver Disease and AUD, MELD-NA Less Than 20 | Alcohol-related Liver Disease and AUD, MELD-NA More Than 20
Started | 6 | 6
Completed | 5 | 2
Not Completed | 1 | 4
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alcohol-related Liver Disease and AUD, MELD-NA Less Than 20 | Alcohol-related Liver Disease and AUD, MELD-NA More Than 20 | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 48 [43.00 to 55.25] | 50 [41.75 to 56.75] | 50 [41.25 to 57.00]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 4 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Adverse Event
Description: Number of adverse events reported
Time Frame: 24 weeks
Population: One MELD-NA less than 20 subject and four MELD-NA more than 20 subjects withdrew prior to initiating the study drug. Data was not collected nor analyzed for those 5 subjects
Measure: Number; unit: adverse events
Arm/Group | Alcohol-related Liver Disease and AUD, MELD-NA Less Than 20 | Alcohol-related Liver Disease and AUD, MELD-NA More Than 20
Number analyzed (Participants) | 5 | 2
adverse events | 0 | 1

2. Secondary Outcome: Change in Alcohol Craving
Description: Number of subjects who experienced a decrease or unchanged Pennsylvania Alcohol Craving Scale (PACS) score from baseline to week 24. Measured using self-reported questionnaire using Pennsylvania Alcohol Craving Scale (PACS). The PACS has 5 questions, where each question has six options presented in Likert Scales from 0 to 6, with 0 being the least and 6 being the highest possible option, thus the possible minimum and maximum values are 0 and 30, respectively. Higher score indicates a positive alcohol craving symptom.
Time Frame: Baseline, week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Alcohol-related Liver Disease and AUD, MELD-NA Less Than 20 | Alcohol-related Liver Disease and AUD, MELD-NA More Than 20
Number analyzed (Participants) | 5 | 2
Participants | 3 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study, approximately 24 weeks.
Arm/Group | Alcohol-related Liver Disease and AUD, MELD-NA Less Than 20 | Alcohol-related Liver Disease and AUD, MELD-NA More Than 20
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alcohol-related Liver Disease and AUD, MELD-NA Less Than 20 (N=6) | Alcohol-related Liver Disease and AUD, MELD-NA More Than 20 (N=6)
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-25): https://cdn.clinicaltrials.gov/large-docs/20/NCT04287920/Prot_SAP_000.pdf